CLINICAL TRIAL: NCT03231865
Title: Diagnostic of Iron Deficiency by Means of Non Invasive Measurement of Zink Protoporphyrin IX
Acronym: ZnPP
Status: Completed | Type: Observational
Sponsor: Philipp Stein (Other)
Responsible Party: Sponsor-Investigator, Philipp Stein, Dr. med Philipp Stein, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2017-00054
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preoperative patients: Patients present themselves before an operation to the Anesthesiologist. They are screened for study eligibility.
  Interventions: Diagnostic Test: Non-invasive measurement of ZincProtoporphyrin IX

INTERVENTIONS:
Diagnostic Test: Non-invasive measurement of ZincProtoporphyrin IX — Within 30 seconds, a measurement is performed on the lip of a patient to determine a ZincProtoporphyrin value

SUMMARY:
ZnPP is being build in the case of a functional iron deficiency. Zinc instead of iron is implemented into protoporphyrin IX. This ZincProtoporphyrin (ZnPP) can be detected non invasively. Non invasive and invasive optical measurement of ZnPP will be compared. Additionally ZnPP measurements will be compared to other iron deficiency parameters for validation by the investigators.

DETAILED DESCRIPTION:
Zinc-protoporphyrin (ZnPP) will be measured by a fluorescence technique. Restricted wave light (407/425 nm) is used to detect ZnPP in the bloodstream non-invasively through the oral mucosa. The spectroscopic measurements are translated into a ZnPP value (mumol/mol heme).

The non-invasive measurement of ZnPP is validated and compared to optical measurement of ZnPP in whole blood and high performance liquid chromatography (HPLC) measurement of ZnPP in whole blood.

The ZnPP value is compared to other iron-deficiency parameters: Ferritin, Transferrin saturation and soluble Transferrin receptor.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen preoperatively in the Anesthestic clinic
* Patients > 18 years of age
* Understood and signed patient consent

Exclusion Criteria:

* transfusion of blood products 8 weeks prior to screening
* Pregnancy
* Porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients prior to a surgery, seen in the Anesthetic clinic for evaluation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Validation of the non-invasive ZincProtoporphyrinIX measurement | Baseline
  The value is compared to optical measurement of ZincProtoporphyrin in whole blood; in addition the value is compared to HPLC measurement in whole blood

SECONDARY OUTCOMES:
Comparison of the ZincProtoporyphyrinIX value to other iron-deficiency parameters | Baseline
  The value is compared to Ferritin, Transferrin saturation and soluble transferrin receptor

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Stein, MD, Principal Investigator — Institute of Anesthesiology, University and University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hennig G, Homann C, Teksan I, Hasbargen U, Hasmuller S, Holdt LM, Khaled N, Sroka R, Stauch T, Stepp H, Vogeser M, Brittenham GM. Non-invasive detection of iron deficiency by fluorescence measurement of erythrocyte zinc protoporphyrin in the lip. Nat Commun. 2016 Feb 17;7:10776. doi: 10.1038/ncomms10776. PMID 26883939